CLINICAL TRIAL: NCT02584218
Title: Effectiveness of Sealing Dental Caries: a Randomized Clinical Trial
Brief Title: Effectiveness of Sealing Dental Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Káiron Ribeiro Dias, Postgraduate student, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGA-0001
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-invasive resin based caries sealing (Experimental): Application of resin based sealant after acid etching of carious occlusal surface
  Interventions: Procedure: Non-invasive resin based caries sealing
- Invasive resin based restoration (Active Comparator): Application of resin based resin restoration after operative intervention of caries lesion, excavation and preparation on occlusal surface
  Interventions: Procedure: Invasive resin based restoration

INTERVENTIONS:
Procedure: Non-invasive resin based caries sealing — The dentists use resin based sealants of own choice, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from The Department of Pediatric Dentistry and Orthodontics, Federal University of Rio de Janeiro, Brazil
  Other Names: Sealing dental caries
  Arms: Non-invasive resin based caries sealing
Procedure: Invasive resin based restoration — The dentists use preparation design and resin composites of own choice, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from The Department of Pediatric Dentistry and Orthodontics, Federal University of Rio de Janeiro, Brazil
  Other Names: Restoration
  Arms: Invasive resin based restoration

SUMMARY:
This study aims to evaluate, through a controlled clinical randomized study, the effectiveness of sealing carious lesions with composite resin in primary molars. For this, healthy children (n=100) with caries lesion reaching to the middle third of the dentin of primary molars, will be submitted to different treatments to remove the lesions. These patients will be randomly allocated in the following treatment groups: (1) cavity sealing (Non-invasive resin based dental sealing) without caries removal; and (2) Partial caries removal and Invasive resin based restoration. The clinical and radiographic success of the treatment groups will be verified by periodic examination of the restorations by USPHS criteria and radiographic subtraction, respectively, which will be checked progression or not of injury. The researcher responsible for these assessments will be blind to the study, whose evaluations will occur after 6, 12, 24 and 36 months of treatment.

DETAILED DESCRIPTION:
The present study will be carried out as a randomized clinical study. Primary, occlusal caries lesions in children, aged 3-8 years old will be treated by non-invasive resin based sealing (n= 50) or resin based restoration (n=50). Randomization between sealing and restoration (1:1) was made by for a resercher at the Federal University of Rio de Janeiro and kept at the clinics in sealed envelopes. The treatments will be examined clinically and radiographically after 6, 12, 24 and 36 years. The treatments are performed and controlled by only one practitioner (the main reseacher of this study) from the Federal University of Rio de Janeiro, Brazil.

Sealing: The dentist will use a resin based sealing, and follow their usual clinical procedures based on the instructions from the manufacturer and the guidelines from the Department of Pediatric Dentistry and Orthodontics of Federal University of Rio de Janeiro, Brazil.

Restoration: The dentist will use preparation design and a resin based resin restoration, and follow their usual clinical procedures (partial caries removal) based on the instructions from the manufacturer and the guidelines from Department of Pediatric Dentistry and Orthodontics of Federal University of Rio de Janeiro, Brazil.

The prevalence of regression, arrest and progression of sealed and restored caries lesions, are computed and related to the clinical and radiological registrations of children, or treatment related factors for assessing of statistically significant correlations.

The influence of each factor on the longevity and need for retreatment of occlusal sealants and restorations, will be assessed using apropriate analyses for statistical treatment of data.

ELIGIBILITY:
Inclusion Criteria:

* Children with good general health; children with caries lesion reaching to the middle third of the dentin of primary molars

Exclusion Criteria:

* Patients with systemic diseases; patient' guardians who did not consent with the study.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of radiographic caries progression in the test group in comparison with the control group | 36 months after the intervention
  Digital bitewing radiographs were taken at baseline and repeated after 6, 12, 24 and 36-months. The radiographical scoring system that will be used is: 1) Regression in depth of lesion (success) 2: Unchanged depth of lesion (success) 3: Progression in depth of lesion (failure)

SECONDARY OUTCOMES:
Longevity of resin composite used as sealants to restore dental caries | 36 months after the intervention
  Clinical evaluation will be performed through clinical examination after 6, 12, 24 and 36-months. The USPHS criteria for evaluating the marginal integrity of the restoration will be used. Clinical scores: Alfa - Restoration showing continuity with the anatomical shape ; Bravo - Restoration discontinuous with the anatomical shape , but the loss of material is not enough to expose the floor of the cavity; Charlie - Restoration discontinuous with the anatomical shape and the loss of material is sufficient to expose the floor of the cavity; and Delta - mobile Restoration fractured or lost.